CLINICAL TRIAL: NCT03228134
Title: Clinical Study on Treatment of Chronic Persistent Bronchial Asthma With Integrated Traditional Chinese and Western Medicine
Brief Title: Clinical Study on Treatment of Chronic Persistent Bronchial Asthma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Longhua Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017LCSY347
Record Dates: First submitted 2017-07-17; First posted 2017-07-24 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Bronchial Asthma
Keywords: treatment； bronchial asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: All treatment group received traditional chinese medicine plus a standard anti-asthma treatment on study entry, and the control group received placebo and standard anti-asthma treatment.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Double-blind trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hanxiao treatment group (Experimental): 80 patients belongs to Hanxiao type of asthma will take Ke Chuan Liu Wei Granule oral therapy twice everyday for 28 days and receive background therapy of ICS and beta2-agonist.
  Interventions: Drug: Ke Chuan Liu Wei Granule
- Hanxiao control group (Sham Comparator): 80 patients belongs to Hanxiao type of asthma will take Ke Chuan Liu Wei Granule placebo oral therapy twice everyday for 28 days and receive background therapy of ICS and beta2-agonist.
  Interventions: Other: Ke Chuan Liu Wei Granule placebo
- Xuxiao treatment group (Experimental): 80 patients of deficiency type of asthma will take Yang He Ping Chuan Granule oral therapy thrice everyday for 28 days and background therapy of ICS and beta2-agonist.
  Interventions: Drug: Yang He Ping Chuan Granule
- Xuxiao control group (Sham Comparator): 80 patients of deficiency type of asthma will take Yang He Ping Chuan Granule placebo oral therapy thrice everyday for 28 days and background therapy of ICS and beta2-agonist.
  Interventions: Other: Yang He Ping Chuan Granule placebo

INTERVENTIONS:
Drug: Ke Chuan Liu Wei Granule — Traditional Chinese Medicine
  Other Names: KCLW Granule
  Arms: Hanxiao treatment group
Drug: Yang He Ping Chuan Granule — Traditional Chinese Medicine
  Other Names: YHPC Granule
  Arms: Xuxiao treatment group
Other: Ke Chuan Liu Wei Granule placebo — Placebo
  Other Names: Placebo
  Arms: Hanxiao control group
Other: Yang He Ping Chuan Granule placebo — Placebo
  Other Names: Placebo
  Arms: Xuxiao control group

SUMMARY:
Investigators aimed to evaluate the clinical efficacy of integrated traditional Chinese and Western medicine in the treatment of asthma, and to further optimize the prescription of Chinese medicine treatment.

DETAILED DESCRIPTION:
The incidence of asthma in China is high and the rate of control is low. Traditional Chinese medicine has a long history of treating asthma, and has a good clinical curative effect.The purpose of this study is to evaluate the clinical efficacy of traditional Chinese medicine in the treatment of asthma, and to further optimize the prescription of Chinese medicine treatment.

In this study, investigators recruited chronic persistent asthma participants, and gave the corresponding western medicine background treatment and traditional Chinese medicine treatment program for 28 days.Participants will undergo a physical examination, lung function, blood and sputum collection.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with chronic persistent asthma
* Patients had positive bronchodilator reversibility test or positive bronchial challenge test or more than 50 parts per billion of FENO before
* Conform to the predetermined 2 TCM Syndrome Types
* Patients who have given written informed consent

Exclusion Criteria:

* Smoking and continuous exposure to hazardous environment
* With fever, or severity of intermittent state, high degree of sustained, or with respiratory failure, etc.
* Pulmonary emphysema, chronic obstructive pulmonary disease, pulmonary emphysema, pulmonary heart disease, pneumonia, lung cancer and other lung diseases
* Patients who are allergic to therapeutic medicine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Asthma control rate change | up to 4 weeks
  Measured the change from Baseline of asthma control rate

SECONDARY OUTCOMES:
Lung function(FEV1, PEF) | Up to 4 weeks
  Measured routine pulmonary ventilation function test
FeNO | Up to 4 weeks
  The fractional concentration of exhaled nitric oxide
Blood routine examination | Up to 4 weeks
  Hematological routine examination
Liver function test | Up to 4 weeks
  Simple liver function test
Cytokine levels of induced sputum | Up to 4 weeks
  Measured cytokine levels of induced sputum supernatant
Kidney function test | Up to 4 weeks
  Simple kidney function test

CONTACTS AND LOCATIONS:
Overall Officials: Huiyong Zhang, Director, Principal Investigator — tcmdoctorzhang@163.com
Locations (5):
- China (5):
  - Fenglin Street Community Health Service Center, Shanghai, Shanghai Municipality
  - Kangjian Street Community Health Service Center, Shanghai, Shanghai Municipality
  - Tianping Street Community Health Service Center, Shanghai, Shanghai Municipality
  - Longhua Hospital Affiliated Shanghai University of TCM, Shanghai, Shanghai Municipality
  - Fengxian District Hospital of TCM, Shanghai, Shanghai Municipality